CLINICAL TRIAL: NCT02879630
Title: Prospective Evaluation of Adjusted Body Weight Dosing of Acyclovir in Obesity
Status: Recruiting | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Aaron Cumpston, PharmD, BCOP, Pharmacy Clinical Specialist, West Virginia University
Other Study IDs: 1501531856
Record Dates: First submitted 2016-08-18; First posted 2016-08-25 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: pharmacokinetics; acyclovir
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obese Patients: Obese patients (patients whose weight is >190% of ideal body weight) will be receive a single dose of I.V. acyclovir sodium 5mg/kg dosed by adjusted body weight as part of their routine care.
- Non-obese Patients: Normal weigh patients (patients whose weight is 80-120% of ideal body weight) will be receive a single dose of I.V. acyclovir sodium 5mg/kg dosed by total body weight as part of their routine care.

SUMMARY:
Patients receiving acyclovir as standard of care will be enrolled into this study. The currently recommended dosing strategy at our institution for obese patients is to receive intravenous acyclovir dosed per an adjusted body weight [IBW + 0.4(TBW-IBW)]. They will have blood drawn once prior to the first dose of acyclovir and 10 times thereafter, over a total time period of 12 hours. These patients will already be hospitalized for other reasons, and will not be required to make additional trips to the hospital. A total of approximately 4-5 tablespoons of blood will be drawn for this study. Ten obese patients and 10 matched control (non-obese) patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Receiving intravenous acyclovir 5 mg/kg (TBW for normal weight patients and ABW40 for obese patients) as part of their routine care
* Weight > 190% of ideal body weight (IBW) for "obese" patients or weight 80-120% of IBW for matched control patients.

Exclusion Criteria:

* Receipt of acyclovir or a pro-drug of acyclovir (valacyclovir, ganciclovir, valganciclovir, famciclovir) in the prior 24 hours
* Serum creatinine >1.5 mg/dL
* Hypersensitivity to acyclovir
* Patients requiring ventilator support or vasopressors in the prior 24 hours
* Receipt of probenecid, mycophenolate, tenofovir, or zidovudine in the prior 7 days
* Significant anatomical deformities that influence body habitus (i.e. amputation)
* Prior inclusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese and non-obese patients receiving intravenous acyclovir
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of systemic acyclovir exposure in obese and non-obese patients | 12 hours

SECONDARY OUTCOMES:
Half-life of acyclovir in obese and non-obese patients | 12 hours
Maximum concentration (Cmax) of acyclovir in obese and non-obese patients | 12 hours
Time to maximum concentration (Tmax) of acyclovir in obese and non-obese patients | 12 hours
Volume of distribution (Vd) of acyclovir in obese and non-obese patients | 12 hours
Systemic Clearance of acyclovir in obese and non-obese patients | 12 hours
Time that concentration is above IC50 for varicella and herpes viruses in obese and non-obese patients | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Cumpston, PharmD, BCOP, Principal Investigator — West Virginia University Medicine
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No